CLINICAL TRIAL: NCT01052077
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of OPDC-34712 (1 to 3 mg/Day) as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder.
Brief Title: Study of the Safety and Efficacy of OPC-34712 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder
Acronym: STEP-D222
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-09-222
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-09

CONDITIONS: Major Depressive Disorder
Keywords: OPC-34712; Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Brexipiprazole + ADT (Experimental): OPC-34712 Tablets, Oral, 1 - 3 mg OPC-34712 + ADT
  Interventions: Drug: OPC-34712; Drug: Placebo; Drug: ADT
- Placebo + ADT (Placebo Comparator): Placebo + ADT
  Interventions: Drug: Placebo; Drug: ADT

INTERVENTIONS:
Drug: OPC-34712 — Tablets, Oral, 1 - 3 mg OPC-34712
  Arms: Brexipiprazole + ADT
Drug: Placebo — Placebo
Drug: ADT
  Other Names: FDA Approved Antidepressant (ADT)

SUMMARY:
This is a Double-blind study wherein patients with Major Depressive Disorder (MDD) will receive either from 1 to 3 mg a day of study medication (OPC-34712)or placebo (an inactive substance) in addition to an FDA approved antidepressant in order to determine if the study medication is effective as an add on treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age, with diagnosis of major depressive disorder, as defined by DSM-IV-TR criteria
* The current depressive episode must be equal to or greater than 8 weeks in duration
* Subjects must report a history for the current depressive episode of an inadequate response to at least one and no more than three adequate antidepressant treatments.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug.
* Subjects who report an inadequate response to more than three adequate trials of antidepressant treatments during current depressive episode at a therapeutic dose for an adequate duration.
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of: Delirium, dementia,amnestic or other cognitive disorder Schizophrenia, schizoaffective disorder, or other psychotic disorder Bipolar I or II disorder
* Subjects with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Southwestern Research, Beverly Hills, California
  - Excell Research, Oceanside, California
  - Affiliated Research Institute, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Clinical InSights, Glen Burnie, Maryland
  - Pharmasite Research, Inc., Pikesville, Maryland
  - MSU/Institute for Health Studies, East Lansing, Michigan
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Northcoast Clinical Trials, Beachwood, Ohio
  - Patient Priority Clinical sites, LLC, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), LLC, Portland, Oregon
  - City Line Avenue Family Practice, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Clinical NeuroScience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Radiant Research, Salt Lake City, Utah
  - Psychiatric Alliance of The Blue Ridge, Charlottesville, Virginia
  - NeuroScience, Inc., Herndon, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin

REFERENCES:
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in the United States in 773 participants at 44 centers. A total of 1226 participants were screened, 773 participants were enrolled in Phase A, and 769 were treated in Phase A. Of the 623 participants who completed Phase A, 372 participants were randomized in to Phase B.
Pre-assignment Details: A 7 to 28-day Screening period, 8-Week single-blind placebo-ADT (antidepressant therapy) prospective Phase, 6-Week double-blind randomization Phase (Phase B), and 30-day follow-up after last dose of medication. Any participant randomized/completed all visits through Week 14 were allowed into an open-label rollover trial (NCT01052077).
Groups:
- Phase A: Participants entered a single-blind prospective treatment phase during which they received single-blind placebo plus open-label commercially available ADT for 8 weeks at maximally tolerated doses.
- Brexiprazole: Participants with an incomplete response at the end of treatment phase (Week 8) were randomized to brexpiprazole arm 1 to 3 mg/day, plus the final dosage of the assigned open-label marketed ADT.
- Placebo: Participants with an incomplete response at the end of treatment phase (Week 8) were randomized to placebo arm plus the final dosage of the assigned open-label marketed ADT.
- Phase A+: Participants who met the criteria for a response at the end of the 8 weeks prospective treatment phase received single-blind placebo + ADT for an additional 6 weeks in Phase A+ for a total of 14 weeks.
Period: Phase A
Arm/Group | Phase A | Brexiprazole | Placebo | Phase A+
Started | 769 | 0 | 0 | 0
Completed | 623 | 0 | 0 | 0
Not Completed | 146 | 0 | 0 | 0
Not completed — Lost to Follow-up | 22 | 0 | 0 | 0
Not completed — Adverse Event | 32 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 26 | 0 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 29 | 0 | 0 | 0
Not completed — Protocol Deviation | 27 | 0 | 0 | 0
Period: Phase B
Arm/Group | Phase A | Brexiprazole | Placebo | Phase A+
Started | 0 | 185 | 187 | 0
Completed | 0 | 167 | 171 | 0
Not Completed | 0 | 18 | 16 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 9 | 2 | 0
Not completed — Met Withdrawal Criteria | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0
Not completed — Protocol Deviation | 0 | 3 | 4 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Period: Phase A+
Arm/Group | Phase A | Brexiprazole | Placebo | Phase A+
Started | 0 | 0 | 0 | 251
Completed | 0 | 0 | 0 | 230
Not Completed | 0 | 0 | 0 | 21
Not completed — Lost to Follow-up | 0 | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 4
Not completed — Met Withdrawal Criteria | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole: Participants with an incomplete response at the end of treatment phase (Week 8) were randomized to brexpiprazole arm 1 to 3 mg/day, plus the final dosage of the assigned open-label marketed ADT.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole | Placebo | Total
Number analyzed (Participants) | 185 | 187 | 372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (11.7) | 42.4 (11.7) | 43.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 130 | 253
  Male | 62 | 57 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change From the End of Phase A (Week 8 Visit) to the End of Phase B (Week 14 Visit) in the Montgomery Asberg Depression Rating Scale (MADRS) Total Score.
Description: The MADRS was utilized as the primary efficacy assessment of a participants level of depression. The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items; therefore, possible total scores range from 0 to 60. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place.
Time Frame: Baseline (end of week 8) to Week 14
Population: The efficacy sample was the Full Analysis Set (FAS) comprised of participants who received 1 dose of double-blind study medication and had both end of Week 8 visit value and 1 post-randomization efficacy assessment for MADRS total score in double-blind Phase B. The LOCF method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
Units on a scale | -8.20 (0.62) | -7.02 (0.62)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.1416, ANCOVA — ANCOVA model, with treatment and study center as main effects and Week 8 value as convariate, is used for change from Week 8 comparisons; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-2.75 to 0.39]

2. Secondary Outcome: Change From End of Phase A (Week 8) to Phase B in Sheehan Disability Scale (SDS) Score.
Description: The SDS was a self-rated instrument used to measure the effect of the participants symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores ranged from 0 through 10. The number most representative of how much each area was disrupted by symptoms was marked along the line from 0= not at all, to 10= extremely. Scores of 5 and above are associated with significant functional impairment. The SDS total score ranges from 0 to 30, with higher values indicating greater disruption in the participant's work/social/family life. For the work/school item, no response was to be entered if the participant did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS score were calculated over the three item scores. All three item scores were needed to be available with the exception of the work/school item score when this item was not applicable.
Time Frame: Baseline (end of week 8) to Week 14
Population: The efficacy sample was the FAS comprised of participants who received 1 dose of double-blind study medication and had both end of Week 8 visit value and 1 post-randomization efficacy assessment for MADRS total score in double-blind Phase B. The LOCF method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 174 | 172
Units on a scale | -0.91 (0.19) | -0.69 (0.19)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.3778, ANCOVA — ANCOVA model, with treatment and study center as main effects and Week 8 value as covariate, is used for change from Week 8 comparisons; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.69 to 0.26]

3. Secondary Outcome: Change From End of Phase A (Week 8 Visit) in MADRS Total Score for Every Trial Week Visit in Phase B.
Description: as for outcome 1
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
Units on a scale
  Week 9 (N= 181, 180) | -3.30 (0.42) | -1.99 (0.42)
  Week 10 (N= 184, 181) | -5.92 (0.50) | -4.01 (0.50)
  Week 11 (N= 184, 181) | -7.23 (0.57) | -5.22 (0.57)
  Week 12 (N= 184, 181) | -8.42 (0.59) | -6.21 (0.59)
  Week 13 (N= 184, 181) | -9.00 (0.59) | -7.18 (0.59)
  Week 14 (N= 184, 181) | -8.20 (0.62) | -7.02 (0.62)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.0162, ANCOVA — ANCOVA model, with treatment and trial center as main effects and Week 8 value as covariate, was used for change from Week 8 comparisons; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.38 to -0.24]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.0031, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-3.15 to -0.65]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0061, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -2.01, 95% CI 2-sided [-3.44 to -0.58]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-3.69 to -0.72]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0174, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-3.32 to -0.32]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.1416, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-2.75 to 0.39]

4. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to Phase B by Study Week in Clinical Global Impression- Severity Illness Scale (CGI-S) Score.
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the investigator had to answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
Units on a scale
  Week 9 (N= 181, 180) | -0.29 (0.05) | -0.20 (0.05)
  Week 10 (N= 184, 181) | -0.58 (0.06) | -0.44 (0.06)
  Week 11 (N= 184, 181) | -0.76 (0.07) | -0.59 (0.07)
  Week 12 (N= 184, 181) | -0.94 (0.07) | -0.68 (0.07)
  Week 13 (N= 184, 181) | -1.00 (0.08) | -0.81 (0.08)
  Week 14 (N= 184, 181) | -0.95 (0.08) | -0.85 (0.08)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.1481, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.21 to 0.03]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.0691, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.28 to 0.01]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0457, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.35 to -0.00]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0061, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.45 to -0.08]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0572, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.38 to 0.01]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.3318, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.29 to 0.10]

5. Secondary Outcome: Change From End of Phase A (Week 8 Visit) to Phase B by Study Week in Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) Total Score.
Description: The IDS-SR was a 30-item self-report measure, that was used to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of major depressive disorder (MDD). For individual items, the scores range from 0 to 3. The IDS-SR are scored by summing responses to 28 of the 30 items to obtain a total score ranging from 0 to 84, higher values indicate greater disruption in the depressive symptoms.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
Units on a scale
  Week 9 (N= 181, 179) | -1.65 (0.54) | -1.99 (0.53)
  Week 10 (N= 184, 181) | -2.91 (0.60) | -2.93 (0.60)
  Week 11 (N= 184, 181) | -3.92 (0.68) | -3.64 (0.68)
  Week 12 (N= 184, 181) | -4.82 (0.74) | -4.76 (0.74)
  Week 13 (N= 184, 181) | -5.60 (0.75) | -5.59 (0.75)
  Week 14 (N= 184, 181) | -5.70 (0.80) | -5.84 (0.80)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.6272, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.02 to 1.69]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.9697, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.48 to 1.54]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.7490, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-2.00 to 1.44]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.9459, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-1.94 to 1.81]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.9893, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-1.91 to 1.88]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.8918, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.89 to 2.17]

6. Secondary Outcome: Change From End of Phase A (Week 8) to End of Phase B (Week 14) in the Hamilton Depression Rating Scale 17-item Version (HAM-D17) Total Score.
Description: The HAM-D17 was utilized as a secondary assessment of a participants level of depression. The HAM-D (17-Item) consisted of 17 items. Eight items were rated on a 0 to 2 scale (items 4, 5, 6, 12, 13, 14, 16 and 17), while nine items (items 1, 2, 3, 7, 8, 9, 10, 11, and 15) were rated on a 0 to 4 scale (twice the weight of the other items). For all of these items, 0 was the "best" rating and the highest score (2 or 4) was the "worst" rating. The possible total scores were from 0 to 52.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 176 | 172
Units on a scale | -5.98 (0.45) | -5.40 (0.45)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.3247, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.71 to 0.57]

7. Secondary Outcome: Clinical Global Impression- Improvement Scale (CGI-I) Score by Study Week in Phase B Relative to End of Phase A.
Description: The efficacy of study medication was rated for each participant using the CGI-I. The study physician would rate the participants total improvement whether or not it is due entirely to drug treatment. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
Units on a scale
  Week 9 (N= 181, 179) | 3.33 (0.82) | 3.37 (0.74)
  Week 10 (N= 184, 180) | 3.03 (0.97) | 3.15 (0.84)
  Week 11 (N= 184, 180) | 3.00 (1.08) | 3.02 (0.99)
  Week 12 (N= 184, 180) | 2.63 (1.12) | 2.91 (1.02)
  Week 13 (N= 184, 180) | 2.60 (1.14) | 2.80 (1.02)
  Week 14 (N= 184, 181) | 2.68 (1.18) | 2.78 (1.07)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.5616, Cochran-Mantel-Haenszel — Cohran-Mantel-Haenszel (CMH) row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean: brexpiprazole - placebo
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.1900, Cochran-Mantel-Haenszel — CMH row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0501, Cochran-Mantel-Haenszel — CMH row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0137, Cochran-Mantel-Haenszel — CMH row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0711, Cochran-Mantel-Haenszel — CMH row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.3438, Cochran-Mantel-Haenszel — CMH row mean scores differ test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo

8. Secondary Outcome: Number of Participants With MADRS Response During Phase B Relative to the End of Phase A (Week 8) Visit.
Description: A MADRS response was defined as >=50 percent reduction in MADRS Total Score from end of Phase A (Week 8 visit). The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items; therefore, possible total scores range from 0 to 60. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
participants
  Week 9 (N= 181, 180) | 11 | 4
  Week 10 (N= 184, 181) | 29 | 16
  Week 11 (N= 184, 181) | 41 | 26
  Week 12 (N= 184, 181) | 56 | 28
  Week 13 (N= 184, 181) | 55 | 33
  Week 14 (N= 184, 181) | 55 | 36
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.0679, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response rate = 2.79, 95% CI 2-sided [0.88 to 8.81]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.0360, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.78, 95% CI 2-sided [1.01 to 3.14]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0521, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.53, 95% CI 2-sided [0.99 to 2.35]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.93, 95% CI 2-sided [1.31 to 2.86]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0074, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.64, 95% CI 2-sided [1.14 to 2.38]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.0339, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.47, 95% CI 2-sided [1.03 to 2.08]

9. Secondary Outcome: Number of Participants With MADRS Remission During Phase B Relative to the End of Phase A (Week 8) Visit.
Description: A MADRS remission was defined as MADRS Total Score =< 10 and >= 50 percent reduction in MADRS Total Score from end of Phase A (Week 8 visit). The MADRS consisted of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS Total Score is the sum of ratings for all 10 items; therefore, possible total scores range from 0 to 60. The MADRS total score were to be unevaluable if less than 8 of the 10 items were recorded. If 8 or 9 of the 10 items were recorded, the MADRS total score was the mean of the recorded items multiplied by 10 and then rounded of to the first decimal place.
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
participants
  Week 9 (N= 181, 180) | 7 | 3
  Week 10 (N= 184, 181) | 15 | 7
  Week 11 (N= 184, 181) | 31 | 18
  Week 12 (N= 184, 181) | 42 | 19
  Week 13 (N= 184, 181) | 46 | 25
  Week 14 (N= 184, 181) | 48 | 27
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.2404, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Remission Rate = 2.27, 95% CI 2-sided [0.55 to 9.30]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.0983, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Remission Rate = 2.04, 95% CI 2-sided [0.83 to 4.98]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0496, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Remission Rate = 1.67, 95% CI 2-sided [0.99 to 2.82]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Remission Rate = 2.12, 95% CI 2-sided [1.31 to 3.46]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0068, Cochran-Mantel-Haenszel; The CMH general association test controlling for trial center; Ratio of Response Rate = 1.77, 95% CI 2-sided [1.17 to 2.67]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.0089, Cochran-Mantel-Haenszel — The CMH general association test controlling for trial center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Ratio of Remission Rate = 1.71, 95% CI 2-sided [1.14 to 2.57]

10. Secondary Outcome: Number of Participants With CGI-Improvement Response During Phase B Relative to the End of Phase A (Week 8).
Description: CGI-I Response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Baseline (end of week 8) to Week 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 184 | 181
participants
  Week 9 (N= 181, 179) | 23 | 19
  Week 10 (N= 184, 180) | 47 | 39
  Week 11 (N= 184, 180) | 73 | 51
  Week 12 (N= 184, 181) | 88 | 63
  Week 13 (N= 184, 181) | 90 | 70
  Week 14 (N= 184, 181) | 84 | 72
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Week 9; Test type: Superiority or Other; p = 0.4605, Cochran-Mantel-Haenszel; CMH general association test controlling for study center; Ratio of Response Rate = 1.23, 95% CI 2-sided [0.70 to 2.18]
Statistical Analysis 2: Comparison: Brexpiprazole vs Placebo; Week 10; Test type: Superiority or Other; p = 0.3267, Cochran-Mantel-Haenszel; CMH general association test controlling for study center; Ratio of Response Rate = 1.20, 95% CI 2-sided [0.83 to 1.72]
Statistical Analysis 3: Comparison: Brexpiprazole vs Placebo; Week 11; Test type: Superiority or Other; p = 0.0230, Cochran-Mantel-Haenszel; CMH general association test controlling for study center; Ratio of Response Rate = 1.37, 95% CI 2-sided [1.05 to 1.80]
Statistical Analysis 4: Comparison: Brexpiprazole vs Placebo; Week 12; Test type: Superiority or Other; p = 0.0105, Cochran-Mantel-Haenszel; CMH general association test controlling for study center; Ratio of Response Rate = 1.36, 95% CI 2-sided [1.08 to 1.71]
Statistical Analysis 5: Comparison: Brexpiprazole vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0417, Cochran-Mantel-Haenszel; CMH general association test controlling for study center; Ratio of Response Rate = 1.26, 95% CI 2-sided [1.01 to 1.58]
Statistical Analysis 6: Comparison: Brexpiprazole vs Placebo; Week 14; Test type: Superiority or Other; p = 0.2345, Cochran-Mantel-Haenszel — CMH general association test controlling for study center; Treatment difference = difference in adjusted mean change: brexpiprazole - placebo; Ratio of Response Rate = 1.15, 95% CI 2-sided [0.91 to 1.44]

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time the participant entered Phase B, throughout the 6-week treatment period (Week 9 to Week 14) and until follow-up at 30 days after the last dose of medication.
Description: SAE was any untoward medical occurrence resulting in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. AE was an exacerbation of an existing problem or a new problem experienced by a participant in a trial, whether or not it was drug related. One participant may have experienced multiple events.
Arm/Group | Brexpiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/185 | 3/187
Other Adverse Events (participants affected / at risk) | 90/185 | 63/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=185) | Placebo (N=187)
Sinus bradycardia (Cardiac disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=185) | Placebo (N=187)
Constipation (Gastrointestinal disorders) | 11 | 4
Diarrhoea (Gastrointestinal disorders) | 10 | 10
Fatigue (General disorders) | 14 | 8
Nasopharyngitis (Infections and infestations) | 12 | 5
Weight increased (Investigations) | 21 | 5
Increased appetite (Metabolism and nutrition disorders) | 14 | 3
Akathisia (Nervous system disorders) | 22 | 9
Insomnia (Psychiatric disorders) | 17 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 10
Headache (Nervous system disorders) | 9 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No